CLINICAL TRIAL: NCT02073006
Title: A Randomised, Double-blind, Placebo-Controlled, Parallel Study to Evaluate the Effects of Lepicol® in Adults With Chronic, Functional Constipation
Brief Title: A Study to Evaluate the Effects of a Natural Supplement in Adults With Chronic Functional Constipation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-048
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Constipation
Keywords: Chronic; Functional; Constipation; less than 3 bowel movements per week
MeSH Terms: conditions — Constipation; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Natural Fibre Supplement (Active Comparator): 2 doses per day for 4 weeks
  Interventions: Dietary Supplement: Natural Fibre Supplement
- Placebo (Placebo Comparator): 2 doses per day for 4 weeks
  Interventions: Dietary Supplement: Natural Fibre Supplement

INTERVENTIONS:
Dietary Supplement: Natural Fibre Supplement — Natural Fibre Supplement 2 doses per day for 4 weeks
  Other Names: Lepicol

SUMMARY:
Constipation is common in the general population, especially in women and in the elderly. Hard stool is a complaint often associated with constipation, which suggests that stool softening would provide a major benefit in the strategy of treatment.

This investigative fibre product is primarily a soluble dietary fibre with added probiotics and a prebiotic. It is not digested in the small intestine and partly remains undigested by bacteria in the gut. Also, as probiotics are believed to help restore a healthy gut flora, reduce pH, assist with digestion of food and reduce gaseous by-products they may aid the improvement of intestinal motility.

The objective of this study is to assess if this investigative, fibre product effects the number of bowel movements per week and if this in turn impacts quality of life and symptoms of constipation.

DETAILED DESCRIPTION:
Constipation is a common condition. Perception of a healthy bowel movement varies widely within and among populations but the Rome III Criteria is a standardised tool that diagnoses functional constipation on the basis of the following symptoms for the last 3 months with symptom onset at least 6 months prior to diagnosis:

1. Must include two or more of the following:

   * Straining during at least 25% of defecations
   * Lumpy or hard stools in at least 25% of defecations
   * Sensation of incomplete evacuation for at least 25% of defecations
   * Sensation of anorectal obstruction/blockage for at least 25% of defecations
   * Manual manoeuvres to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor)
   * Fewer than three defecations per week
2. Loose stools are rarely present without the use of laxatives
3. Insufficient criteria for irritable bowel syndrome

Additional to being extremely uncomfortable, untreated constipation can lead to faecal impaction (with resulting faecal incontinence), particularly in elderly and confused people and is believed to be a risk factor for haemorrhoids (piles) and diverticular disease. However even without a medical diagnosis the undesired symptoms can reduce perceived quality of life and successful management may involve a number of factors. Standard treatment consists of disimpaction and the administration of laxatives to achieve a normal bowel habit of passing a soft stool without pain. The daily use of laxatives long term is often advised against as it can make your body dependent on them, causing your bowel to no longer function normally.

Stool softening is a physician's first step in the management of chronic constipation. Psyllium has been shown to soften stools by increasing stool water content, far more than most common dietary fibres. It forms a soft gel which eases the stool along the lower digestive tract ready for evacuation. This bulkier faeces presses on the wall of the intestine, stimulating the muscles to contract and force the contents forward, a process known as 'peristalsis'. If there is insufficient fibre in the diet, the faeces will move more slowly and there will be more time for water to be absorbed from the ingested food into the rest of the body, leaving the faeces smaller and harder, which in turn is more difficult to move. Psyllium has the advantage of being much gentler than some common fibres (such as wheat bran) that can be irritating to a sensitive bowel.

Studies using psyllium in a range of doses of 7g up to 24g a day show positive results in relation to increasing stool frequency and weight, and improving stool consistency, in turn improving associated abdominal pain and discomfort. These results were applicable in both adults and the elderly. Although psyllium works in a much more gentle natural way, in some studies it was seen to be superior to or comparative to commonly used laxatives.

Probiotics had the added advantage of improving stool frequency and consistency and accompanying abdominal pain, most likely by their positive effects on the gut microflora often seen to be imbalanced in those with constipation. These effects were seen in infants, adults and the elderly with no adverse events such inducing loose stools.

Lastly, inulin in a range of doses of 1.5g up to 50g a day was seen to improve not only beneficial bacteria counts but also bowel transit in infants, adults and the elderly and in one study was again seen to be more effective than a common laxative but without the side effects.

This study aims to increase the body of scientific data on psyllium by way of a randomised, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

1. Be able to give written informed consent,
2. Be between 18 and 80 years of age,
3. Subject has chronic functional constipation according to the Rome III Diagnostic Criteria, where (f) is mandatory.

   i. Must include two or more of the following:
   1. Straining during at least 25% of defæcations
   2. Lumpy or hard stools in at least 25% of defæcations
   3. Sensation of incomplete evacuation for at least 25% of defæcations
   4. Sensation of anorectal obstruction / blockage for at least 25% of defaecations
   5. Manual manœuvers to facilitate at least 25% of defæcations (e.g., digital evacuation, support of the pelvic floor)
   6. Fewer than 3 defæcations per week ii. Loose stools are rarely present without the use of laxatives iii. Insufficient criteria for irritable bowel syndrome * Criteria fulfilled for the last 3 months, with symptom onset at least 6 months prior to diagnosis
4. Subjects will continue on his/her normal diet,
5. The subject agrees to complete the Patient Diary for two weeks prior to study entry and for the duration of the study.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Are less than 18 and greater than 80 years of age,
2. Females are pregnant, lactating or wish to become pregnant during the study.
3. Are hypersensitive to any of the components of the test product,
4. Have a significant acute or chronic, unstable and untreated disease or any condition which contraindicates, in the investigators judgement, entry to the study,
5. Subject has an obstructive or metabolic aetiology for constipation,
6. Subject has a history of laxative abuse (greater than the daily dosage recommended on the label for any laxative),
7. Subject has used a probiotic or prebiotic product or a dietary fibre supplement in the 4 weeks prior to the baseline visit,
8. Subject has a history of drug and/or alcohol abuse at the time of enrolment
9. Having a condition or have taken a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results;
10. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial,
11. Subjects may not be receiving treatment involving experimental drugs,
12. If the subject has been in a recent experimental trial, these must have been completed not less than 90 days prior to this study.
13. Have a malignant disease or any concomitant end-stage organ disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of bowel movements per week | 4 weeks

SECONDARY OUTCOMES:
Stool consistency, as measured by the Bristol Stool Form Scale | 4 weeks
Quality of life as measured by the Quality of Life Questionnaire (PAC-QOL) | 4 weeks
Constipation symptoms as measured by PAC-SYM | 4 weeks
Laxative use by subjects with functional constipation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, MD,FRCP,FACG, Principal Investigator — Cork University Hospital
Locations (1):
- Atlantia Food Clinical Trials, University College Cork, Cork, Ireland